CLINICAL TRIAL: NCT01593267
Title: Barrow Ruptured Aneurysm Study
Brief Title: Barrow Ruptured Aneurysm Trial
Acronym: BRAT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. Joseph's Hospital and Medical Center, Phoenix (Other)
Collaborators: Barrow Neurological Foundation (Other); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Lisa Arnold, Research Operations Manager, St. Joseph's Hospital and Medical Center, Phoenix
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02BN090
Record Dates: First submitted 2012-04-30; First posted 2012-05-08 (Estimated); Last update posted 2021-09-21 (Actual); Status verified 2021-09

CONDITIONS: Ruptured Cerebral Aneurysm; Subarachnoid Hemorrhage (SAH)
Keywords: intracranial aneurysm; subarachnoid hemorrhage; randomized trial; coil embolization; clip occlusion; vascular disorders
MeSH Terms: conditions — Subarachnoid Hemorrhage; Intracranial Aneurysm; Vascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endovascular (Active Comparator): Subjects randomized to endovascular coil embolization will be treated by one of two neurosurgeons expert in such treatment. All endovascular coil embolization treatments will be accomplished using accepted techniques.
  Interventions: Procedure: coil embolization
- Surgical (Active Comparator): Subjects randomized to surgical clip occlusion repair will receive treatment from one of two neurosurgeons expert in clip occlusion surgery for ruptured aneurysms.
  Interventions: Procedure: clip occlusion

INTERVENTIONS:
Procedure: coil embolization — Subjects randomized to endovascular therapy will be treated by one of two neurosurgeons expert in such treatment. All endovascular treatments will be accomplished using accepted techniques.
  Arms: Endovascular
Procedure: clip occlusion — Subjects randomized to surgical therapy will receive treatment from one of two neurosurgeons expert in surgery for ruptured aneurysms.
  Arms: Surgical

SUMMARY:
With evolving endovascular technologies there is a growing debate centered on the relative safety and efficacy of the currently accepted alternatives for the treatment of ruptured cerebral aneurysms in the face of acute subarachnoid hemorrhage (SAH). The purpose of this study is to compare the safety and efficacy of microsurgical clipping and endovascular coiling of acutely ruptured cerebral aneurysms in a prospective, randomized fashion.

DETAILED DESCRIPTION:
The planned trial enrolled 250 subjects per arm. Subjects are followed postoperatively and outcome endpoints will be assessed at Discharge, 6 Months, 1 Year, 3 Years, and 6 Years. One hundred (100) subjects will participate in neuropsychological testing at 1 Year; after the 100th subject an interim data analysis will be performed and the viability of future neuropsychological testing will be determined. Subjects will receive preoperative, intraoperative or postoperative, 3 Year follow up, and 6 Year follow up angiograms. In this fashion immediate clinical outcome, including peri-procedural morbidity and mortality, will be assessed as will long term outcome, both clinical and angiographic.

ELIGIBILITY:
Inclusion Criteria:

* Acute subarachnoid hemorrhage (SAH)
* Confirmed by CT scan or lumbar puncture
* Age 18-80 years
* Ability to give informed consent (subject or legally authorized representative)
* No anatomic inclusions

Exclusion Criteria:

* Traumatic subarachnoid hemorrhage
* Presents to hospital >14 days post-bleed
* SAH caused by other primary disease
* No anatomic exclusions

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2002-11; Primary Completion 2019-10-25 (Actual); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Modified Rankin Scale | 10 years
  Primary Outcome Measure is Modified Rankin Scale < or = to 2. Data will be analyzed on intent to treat basis with crossover to the alternative treatment analyzed as a data subset. The null hypothesis is that no difference in outcome will be detected between the endovascular and surgical treatment arms. A statistically significant difference will then be considered evidence in favor of the alternative hypothesis, that one treatment is superior to the other.

CONTACTS AND LOCATIONS:
Overall Officials: Robert F Spetzler, MD, Principal Investigator — Barrow Brain and Spine
Locations (1):
- St. Joseph's Hospital and Medical Center, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Catapano JS, Zabramski JM, Baranoski JF, Brigeman S, Morgan CD, Hendricks BK, Mooney MA, Albuquerque FC, Nakaji P, Spetzler RF. The Prognostic Significance of a Cast Fourth Ventricle in Ruptured Aneurysm Patients With Intraventricular Hemorrhage in the Barrow Ruptured Aneurysm Trial (BRAT). Neurosurgery. 2019 Aug 1;85(2):E275-E283. doi: 10.1093/neuros/nyy493. PMID 30476225
- [Background] Mascitelli JR, Lawton MT, Hendricks BK, Nakaji P, Zabramski JM, Spetzler RF. Analysis of Wide-Neck Aneurysms in the Barrow Ruptured Aneurysm Trial. Neurosurgery. 2019 Nov 1;85(5):622-631. doi: 10.1093/neuros/nyy439. PMID 30346618
- [Background] Mooney MA, Simon ED, Brigeman S, Nakaji P, Zabramski JM, Lawton MT, Spetzler RF. Long-term results of middle cerebral artery aneurysm clipping in the Barrow Ruptured Aneurysm Trial. J Neurosurg. 2019 Mar 1;130(3):895-901. doi: 10.3171/2017.10.JNS172183. Epub 2018 Apr 27. PMID 29701554
- [Background] Mooney MA, Brigeman S, Bohl MA, Simon ED, Sheehy JP, Chang SW, Spetzler RF. Analysis of overlapping surgery in patients undergoing microsurgical aneurysm clipping: acute and long-term outcomes from the Barrow Ruptured Aneurysm Trial. J Neurosurg. 2018 Sep;129(3):711-717. doi: 10.3171/2017.5.JNS17394. Epub 2017 Nov 3. PMID 29099301
- [Background] Spetzler RF, Zabramski JM, McDougall CG, Albuquerque FC, Hills NK, Wallace RC, Nakaji P. Analysis of saccular aneurysms in the Barrow Ruptured Aneurysm Trial. J Neurosurg. 2018 Jan;128(1):120-125. doi: 10.3171/2016.9.JNS161301. Epub 2017 Feb 24. PMID 28298031
- [Background] McDougall CG, Spetzler RF, Albuquerque FC, Zabramski JM, Nakaji P. Crossover and clinical outcomes in the Barrow Ruptured Aneurysm Trial. Response. J Neurosurg. 2014 Feb;120(2):572. No abstract available. PMID 24645176
- [Result] McDougall CG, Spetzler RF, Zabramski JM, Partovi S, Hills NK, Nakaji P, Albuquerque FC. The Barrow Ruptured Aneurysm Trial. J Neurosurg. 2012 Jan;116(1):135-44. doi: 10.3171/2011.8.JNS101767. Epub 2011 Nov 4. PMID 22054213
- [Result] Spetzler RF, McDougall CG, Albuquerque FC, Zabramski JM, Hills NK, Partovi S, Nakaji P, Wallace RC. The Barrow Ruptured Aneurysm Trial: 3-year results. J Neurosurg. 2013 Jul;119(1):146-57. doi: 10.3171/2013.3.JNS12683. Epub 2013 Apr 26. PMID 23621600
- [Result] Spetzler RF, McDougall CG, Zabramski JM, Albuquerque FC, Hills NK, Nakaji P, Karis JP, Wallace RC. Ten-year analysis of saccular aneurysms in the Barrow Ruptured Aneurysm Trial. J Neurosurg. 2019 Mar 8;132(3):771-776. doi: 10.3171/2018.8.JNS181846. Print 2020 Mar 1. PMID 30849758
- [Result] Mascitelli JR, Cole T, Yoon S, Nakaji P, Albuquerque FC, McDougall CG, Zabramski JM, Lawton MT, Spetzler RF. External Validation of the Subarachnoid Hemorrhage International Trialists (SAHIT) Predictive Model Using the Barrow Ruptured Aneurysm Trial (BRAT) Cohort. Neurosurgery. 2020 Jan 1;86(1):101-106. doi: 10.1093/neuros/nyy600. PMID 30566611
- [Result] Spetzler RF, McDougall CG, Zabramski JM, Albuquerque FC, Hills NK, Russin JJ, Partovi S, Nakaji P, Wallace RC. The Barrow Ruptured Aneurysm Trial: 6-year results. J Neurosurg. 2015 Sep;123(3):609-17. doi: 10.3171/2014.9.JNS141749. Epub 2015 Jun 26. PMID 26115467
- [Derived] Labib MA, Catapano JS, Inoue M, Kupanoff KM, Singh R, Abramov I, Scherschinski L, Srinivasan VM, Youn TS, Spetzler RF, Lawton MT. External Validation of the Modified Southwestern Aneurysm Severity Index in the Barrow Ruptured Aneurysm Trial Surgical Cohort. Neurosurgery. 2024 Sep 1;95(3):660-668. doi: 10.1227/neu.0000000000002959. Epub 2024 Apr 29. PMID 38682903